CLINICAL TRIAL: NCT00563537
Title: Molecular Imaging Modality by Positron Emission Tomography Using 18F-X : Study of Microglial Activation in Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: University Hospital, Tours
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRC05-PC / SLA
Record Dates: First submitted 2007-11-22; First posted 2007-11-26 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Bulbar Disease; Spinal Disease
Keywords: neurology; sclerosis; imaging; tomography
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Spinal Diseases; Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 18F-X PET Scan imaging
  Interventions: Radiation: 18F-X PET SCAN

INTERVENTIONS:
Radiation: 18F-X PET SCAN — 18F-X PET Scan : Injection of 7.8 mSv for 370 MBq of dose (0.021 mSv / MBq)

SUMMARY:
PET imaging of activated microglia offers a tool of investigation of a range of brain diseases where neuroinflammation is a component.

Amyotrophic lateral sclerosis is the most frequent motoneuronal disease in adult.

This study was designed to explore the feasibility of molecular imaging modality by Positron Emission Tomography using 18F-X as an in vivo marker of activated microglia for the assessment of neuroinflammation in amyotrophic lateral sclerosis.

PET may help in the diagnosis of the disease and, further, may allow assessment of the efficacy of antiinflammatory treatment.

DETAILED DESCRIPTION:
18F-X PET will be carried out requiring arterial sampling in 2 patients suffering from ALS and 2 normal subjects in order to evaluate the 18F-X quantification.

Then simplified PET using 18F-X will be carried out in 13 patients and 13 normal subjects.

Binding potential maps showing specific binding of 18f-X will be generated for each subject.

Regional binding potential values will be calculated for anatomically defined regions of interest after coregistration to and special transformation into the subject's own MRI.

ELIGIBILITY:
Inclusion Criteria:

* suffering from probable or definite form of amyotrophic lateral sclerosis according to El Escorial criteria. Spinal or bulbar site of the disease.
* Information and signature of the written consent form
* French Social Security registration

Exclusion Criteria:

* family history of ALS
* Riluzole treatment before the first PETscan.
* Psychiatric disorders
* Evolution of the disease older than 18 months
* Antiinflammatory or antibiotic treatment in the last month

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-01; Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative in vivo-imaging of 18F-X microglial binding site as a mesure of disease activity followed up by non invasive quantification of patients using imaging modality. | Inclusion period

SECONDARY OUTCOMES:
Evidence of the localisation of benzodiazepine binding site related to microglial activation in ALS | inclusion period
Evidence of the difference of microglial localisation and activation between bulbar and spinal form of amyotrophic lateral sclerosis | inclusion period

CONTACTS AND LOCATIONS:
Overall Officials: Denis GUILLOTEAU, PHD, Study Director — Service de médecine nucléaire in Vitro - CHRU TOURS; Philippe CORCIA, MD, Principal Investigator — Service de Neurologie - CHRU Tours
Locations (1):
- Service de Médecine Nucléaire et Ultrasons - Hôpital Bretonneau, Tours, Centre-Val de Loire, France

REFERENCES:
- [Background] Kassiou M, Meikle SR, Banati RB. Ligands for peripheral benzodiazepine binding sites in glial cells. Brain Res Brain Res Rev. 2005 Apr;48(2):207-10. doi: 10.1016/j.brainresrev.2004.12.010. Epub 2005 Jan 22. PMID 15850659
- [Background] Banati RB. Visualising microglial activation in vivo. Glia. 2002 Nov;40(2):206-217. doi: 10.1002/glia.10144. PMID 12379908
- [Result] Banati RB, Newcombe J, Gunn RN, Cagnin A, Turkheimer F, Heppner F, Price G, Wegner F, Giovannoni G, Miller DH, Perkin GD, Smith T, Hewson AK, Bydder G, Kreutzberg GW, Jones T, Cuzner ML, Myers R. The peripheral benzodiazepine binding site in the brain in multiple sclerosis: quantitative in vivo imaging of microglia as a measure of disease activity. Brain. 2000 Nov;123 ( Pt 11):2321-37. doi: 10.1093/brain/123.11.2321. PMID 11050032
- [Result] Zhang MR, Kumata K, Maeda J, Yanamoto K, Hatori A, Okada M, Higuchi M, Obayashi S, Suhara T, Suzuki K. 11C-AC-5216: a novel PET ligand for peripheral benzodiazepine receptors in the primate brain. J Nucl Med. 2007 Nov;48(11):1853-61. doi: 10.2967/jnumed.107.043505. PMID 17978354
- [Result] Zhang MR, Maeda J, Ogawa M, Noguchi J, Ito T, Yoshida Y, Okauchi T, Obayashi S, Suhara T, Suzuki K. Development of a new radioligand, N-(5-fluoro-2-phenoxyphenyl)-N-(2-[18F]fluoroethyl-5-methoxybenzyl)acetamide, for pet imaging of peripheral benzodiazepine receptor in primate brain. J Med Chem. 2004 Apr 22;47(9):2228-35. doi: 10.1021/jm0304919. PMID 15084121
- [Derived] Corcia P, Tauber C, Vercoullie J, Arlicot N, Prunier C, Praline J, Nicolas G, Venel Y, Hommet C, Baulieu JL, Cottier JP, Roussel C, Kassiou M, Guilloteau D, Ribeiro MJ. Molecular imaging of microglial activation in amyotrophic lateral sclerosis. PLoS One. 2012;7(12):e52941. doi: 10.1371/journal.pone.0052941. Epub 2012 Dec 31. PMID 23300829